CLINICAL TRIAL: NCT05321628
Title: Evaluating the Effect of Different Clinical Routines and Supervision for ICBT
Brief Title: Evaluating Clinical Routines for ICBT
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Karolinska Institutet (Other)
Collaborators: Region Stockholm (Other Government)
Responsible Party: Principal Investigator, Viktor Kaldo, Clinical Professor, Karolinska Institutet
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 2020-05772
Record Dates: First submitted 2022-03-18; First posted 2022-04-11 (Actual); Last update posted 2025-01-17 (Actual); Status verified 2025-01

CONDITIONS: Depression; Panic Disorder; Social Anxiety Disorder
Keywords: Internet treatment; cognitive behavioral therapy; clinical decision support tool
MeSH Terms: conditions — Depression; Panic Disorder; Phobia, Social

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Masking Description: The therapists and patients will know that they are randomized, but will be informed that the randomization concerns two different types of clinical routines and supervision, and will thus be blind to the true purpose of randomization. Outcome assessors will not be informed that any randomization has occurred.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- iCBT + Decision Support Tool (Experimental): Internet-based Cognitive Behavioural Therapy where therapists have traditional clinical routines and supervision and also use a clinical decision support tool.
  Interventions: Behavioral: Internet-based Cognitive Behavioural Therapy (iCBT) with Decision Support Tool
- Traditional iCBT (Active Comparator): Internet-based Cognitive Behavioural Therapy with traditional clinical routines and supervision.
  Interventions: Behavioral: Internet-based Cognitive Behavioural Therapy (iCBT)

INTERVENTIONS:
Behavioral: Internet-based Cognitive Behavioural Therapy (iCBT) with Decision Support Tool — Cognitive Behavioural Therapy för depression, panic disorder and social anxiety delivered thru texts and home works assignments via an internet platform with therapist weekly support through text messages. Therapist use a traditional, detailed therapist manual with the additions of a Clinical Decision Support Tool (DST) that identifies patients at risk of treatment failure and give suggestions to the therapist on how to act in relation to the specific patient.
  Arms: iCBT + Decision Support Tool
Behavioral: Internet-based Cognitive Behavioural Therapy (iCBT) — iCBT, as described above, using only the traditional, detailed therapist manual.
  Arms: Traditional iCBT

SUMMARY:
The overall aim of this study is to test the clinical benefits of an AI-based decision support tool (DST) and to evaluate how the DST affects therapists and their patients with depression, social anxiety, or panic disorder during 12 weeks of ICBT.

DETAILED DESCRIPTION:
The project aims to evaluate if therapist-supported ICBT with a DST that guides therapists in addition to a traditional therapist manual (the DST arm) are superior to ICBT using only the therapist manual (TRAD) arm.

The investigators hypothesize that DST, in comparison to TRAD, will:

* decrease the diagnose-specific symptoms during the treatment period, among patients identified to be at risk of failure (primary outcome),
* decrease the number of failed treatments among patients identified to be at risk,
* improve everyday functioning, health related quality of life, patient satisfaction, number of Adverse Events experienced by the patient, need for further treatment and sudden symptom changes among patients at risk,
* Increase the therapists' amount of interaction and time spent on patients at risk,
* increase the adherence to treatment among patients at risk, and
* improve levels of symptoms, functioning, interaction, and adherence when all patients (also those not at risk) are included
* make therapists overall more time efficient, defined as the ratio of 'decrease in symptoms / therapist time spent on patient'
* increase therapist experience of using the DST / the therapist manual, including higher perceived helpfulness and credibility and the overall experience of supervision, clinical routines, and guidance of their clinical decisions

The study is designed as a triple blind randomized controlled trial, where half of the therapists are allocated to DST and the other half to TRAD. Each patient is also randomized between those conditions. The therapists and patients will be blind to what group they are allocated to and the post-treatment assessors will also be blind to what group the patients belong to. The therapists and patients will know that they are randomized, but will be informed that the randomization concerns two different types of clinical routines and supervision, and will thus be blind to the true purpose of randomization. After randomization both groups will be informed that they are in the experimental group to lower the risk for nocebo effects.

The DST provides visual feedback about patient current adherence and symptoms levels, as well as predictions of final outcome and adherence, and also use four color indicators to guide the therapist:

* Green: Patient likely to succeed, consider spending less time on patient.
* Yellow: Prediction too uncertain to give guidance.
* Light Red: Patient likely to fail, consider adjustments.
* Dark Red: Patient very likely to fail, adjustments must be implemented.

A patient is considered to be at risk to fail if he/she gets a Light Red or Dark Red indication.

Primary outcome is the diagnose-specific symptom rating for each of the three ICBT-treatments that are used in the trial for Depression (MADRS-S), Panic Disorder (PDSS-SR), and Social Anxiety Disorder (LSAS-SR) respectively. Failed treatment are defined as being neither a responder (50% symptom reduction) nor a remitter (under a previously specified cut-off for each respective diagnose-specific symptom measure).

Primary analyses are performed according to intent-to-treat and, to handle missing data, with an HLM-model that test the interaction of Time x Arm and includes all available symptom data from pre to post, including weekly measures during treatment. It includes the estimated 50% of all patients that will be indicated as at risk (i.e. also control patients in TRAD, although their therapists never see the prediction because they do not use the DST). In a previous proof-of-concept trial the effect corresponding to our primary analysis was Cohen's d=0.59. To be conservative it was estimated to be 0.50. A power of 80% and an attrition of 20% would require 158 patients identified as at risk of failure, and thus 316 in total. To increase the less easily estimated power for secondary measures, the aim is to include 350 patients.

The trial will follow the guidelines of Good Clinical Practice adapted for psychological treatment.

ELIGIBILITY:
Inclusion Criteria:

* 18 years or older.
* Social anxiety, panic disorder or depression diagnosis.
* Stable or no antidepressant medication for at least 2 months.
* No diseases, disorders, or substance abuse that required other, immediate attention (e.g., severe depression or suicidality).
* Available time for treatment and acceptance of its format.
* Proficient in Swedish.
* No ongoing CBT.

Exclusion Criteria:

* Not available for assessment and diagnostic telephone interview.
* Will not be in Sweden during the treatment period.
* Not able to receive text messages on a Swedish mobile phone.
* Not proficient in Swedish.
* No access to computer and internet.
* Not able to set aside about one hour a day to work on treatment.
* Bipolar disorder, if seeking depression treatment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 401 (Actual)
Dates: Start 2021-12-03 (Actual); Primary Completion 2024-10-03 (Actual); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Montgomery-Åsberg Depression Rating Scale-Self report version (MADRS-S) | Measured at pre-treatment, each week in treatment, post (12 weeks after pre), and follow-up after 1 year. Primary endpoint is difference in change/slope during treatment, based on available data from pre-treatment, weekly measures and post-treatment.
  A self-rating scale for depression, specially developed to be sensitive to change. Is in this study the primary symptom measure for depression, where higher scores means more symptoms of depression. Min - Max score = 0 - 54
Panic Disorder Severity Scale - Self Rated (PDSS-SR) | Measured at pre-treatment, each week in treatment, post (12 weeks after pre), and follow-up after 1 year. Primary endpoint is difference in change/slope during treatment, based on available data from pre-treatment, weekly measures and post-treatment.
  A self-report scale for panic disorder that has been shown to be sensitive to change with treatment. Is in this study the primary symptom measure for panic disorder, where higher scores means more panic disorder symptoms. Min - Max score = 0 - 28
Liebowitz Social Anxiety Scale, self-report (LSAS-SR) | Measured at pre-treatment, each week in treatment, post (12 weeks after pre), and follow-up after 1 year. Primary endpoint is difference in change/slope during treatment, based on available data from pre-treatment, weekly measures and post-treatment.
  A self-rated scale for assessment of social anxiety disorder and it has two subscales for fear and avoidance. Is in this study the primary symptom measure for social anxiety, where higher scores means more symptoms of social anxiety. Min - Max score = 0 - 144

SECONDARY OUTCOMES:
Failed/Successful Treatment | From pre-treatment to post-treatment (12 weeks after pre). Sensitivity analysis: to post (12 weeks after pre) or last available weekly symptom measure
  Failure are defined as being neither a responder (50% symptom reduction from pre-treatment) nor a remitter (<11 on MADRS-S; <8 on PDSS-SR; or <36 on LSAS-SR)
Euroqol (EQ-5D) | Screening, post-treatment (12 weeks after pre) and follow-up after 1 year.
  A short questionnaire for measuring health related quality of life.
WHO Disability Assessment Schedule (WHODAS) | Screening, post-treatment (12 weeks after pre) and follow-up after 1 year.
  A self-rated measure of daily functioning and an assessment instrument for health and disability available in 36- and 12-item versions. We will use the 12-item version (WHODAS-12).
Treatment adherence questionnaire | Tri-weekly during treatment and at post-treatment (12 weeks after pre).
  Questions focusing on how they patients have worked with the treatment.
Internet Psychiatry Clinic evaluation questionnaire (version 3). | Post-treatment (12 weeks after pre)
  Client Satisfaction Questionnaire 8 items version (CSQ-8) + 18 items concerning patients experience of the treatment in general, the treatment program, and adverse events.
Patient experience | Post-treatment (12 weeks after pre)
  Specifically designed questions focusing on patients experience of the treatment adaptations, feelings of empowerment, and other aspects of treatment.
Treatment Credibility | Week 3 in treatment
  Patient-rated Treatment Credibility Scale (min - max = 0 - 50, higher scores indicate higher perceived treatment credibility)
Adverse Events | At post-treatment (12 weeks after pre)
  Number of Adverse Events and Serious Adverse Events reported by patient
Need for further treatment | At post-treatment (12 weeks after pre)
  Patient reported need for further treatment

OTHER OUTCOMES:
Time spent by therapist on each patient. | At each interaction with patient and post-treatment (12 weeks after pre).
  Logged in the treatment plattform.
Number of treatment modules each patient has completed. | Throughout treatment from pre-treatment to post (12 weeks after pre)
  Coded from the treatment plattform.
Time efficiency | Throughout treatment from pre-treatment to post (12 weeks after pre)
  Degree of change on primary outcome divided by therapist time spent on the patient.
Therapist experience of using DST / manual (not related to a specific patient) | Time-point not possible to specify in weeks. Measured either when the therapist has fully treated 5 patients or when the therapist leave the study (if that happens before treating 5 patients and has treated at least 1 patient)
  Therapists experience of using the DST / the therapist manual, including perceived helpfulness and credibility and the overall experience of supervision, clinical routines, and guidance of their clinical decisions.
System Usability Scale (SUS) | Time-point not possible to specify in weeks. Measured either when the therapist has fully treated 5 patients or when the therapist leave the study (if that happens before treating 5 patients and has treated at least 1 patient)
  Measuring usability of the DST from the therapist perspective (not related to a specific patient). Min - Max score = 10 - 50

CONTACTS AND LOCATIONS:
Overall Officials: Viktor Kaldo, Principal Investigator — Karolinska Institutet
Locations (1):
- Internet Psychiatry Unit, Psykiatri Sydväst, SLSO, Stockholm, Huddinge, Sweden